CLINICAL TRIAL: NCT06752291
Title: EFFECTIVENESS of WATER FLOSS in PLAQUE REMOVAL and PREVENTION of WHITE SPOT LESIONS in ORTHODONTIC PATIENTS: a RANDOMISED CONTROLLED CLINICAL TRIAL
Acronym: WATER FLOSS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Afif Shafie bin Abd Samad, DR, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DF CD 2424/0060 (P); UMG052E-2024 (Other Grant/Funding Number: UNIVERSITI MALAYA)
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-04

CONDITIONS: White Spot Lesion of Tooth; Gingival Inflammation; Gingival Bleeding; Dental Plaque
Keywords: water flosser; white spot lesion
MeSH Terms: conditions — Gingivitis; Gingival Hemorrhage; Dental Plaque

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Groups of orthodontic patients with experimental interdental cleaning tools ( Water Flosser ) (Experimental): Groups of orthodontic patients with Water Flosser
  Interventions: Device: water flosser
- Groups of orthodontic patients with controlled interdental cleaning tools (No Intervention): Groups of orthodontic patients with controlled interdental cleaning tools ( dental floss and interdental brush)

INTERVENTIONS:
Device: water flosser — A water flosser will be provided for use throughout the study, with participants instructed to use it once daily, specifically at the end of the day before bedtime.
  Arms: Groups of orthodontic patients with experimental interdental cleaning tools ( Water Flosser )

SUMMARY:
This clinical trial aims to learn if water floss is as efficient as other interdental cleaning tools and can prevent plaque accumulation and white spot lesions (WSLs) in orthodontic patients. It will also assess the impact of water floss on gingival health. The main questions it aims to answer are:

* Which interdental cleaning tools reduce plaque accumulation and improve gingival health in orthodontic patients?
* Which interdental cleaning tools lower the incidence of white spot lesions compared to conventional oral hygiene practices? Researchers will compare the oral health of Orthodontic patients' using different interdental cleaning tools to evaluate their effectiveness in improving oral health outcomes.

Participants will:

* Be assigned to one of two groups:

  * Intervention group: instructed to use water flossing in their oral hygiene routine.
  * Control group: instructed to use dental floss and interdental brush in their oral hygiene routine.
* Participate for 8 months, with clinical assessments for plaque and gingival health and photographic documentation for WSLs at baseline (T0), and at 2-month intervals (T1, T2, T3, and T4).

DETAILED DESCRIPTION:
This clinical trial aims to learn if water floss is as efficient as other interdental cleaning tools and can prevent plaque accumulation and white spot lesions (WSLs) in orthodontic patients. It will also assess the impact of water floss on gingival health. The main questions it aims to answer are:

* Which interdental cleaning tools reduce plaque accumulation and improve gingival health in orthodontic patients?
* Which interdental cleaning tools lower the incidence of white spot lesions compared to conventional oral hygiene practices? Researchers will compare the oral health of Orthodontic patients' using different interdental cleaning tools to evaluate their effectiveness in improving oral health outcomes.

Participants will:

* Be assigned to one of two groups:

  * Intervention group: instructed to use water flossing in their oral hygiene routine.
  * Control group: instructed to use dental floss and interdental brush in their oral hygiene routine.
* Participate for 8 months, with clinical assessments for plaque and gingival health and photographic documentation for WSLs at baseline (T0), and at 2-month intervals (T1, T2, T3, and T4).

Aim of the study:

To evaluate the effectiveness of Water Floss in plaque removal and preventing WSLs among orthodontic patients.

Primary Objectives

1. To measure the effectiveness of the water floss in plaque removal based on the Oral Plaque Index (OPI) among fixed appliance patients at T0, T1, T2, T3, and T4.
2. To measure the effectiveness of water flosser based on the incidence of White Spot Lesions (WSLs) among fixed appliance patients at 0 months (T0), 3 months (T1), 6 months (T2), 9 months (T3), and 12 months (T4).
3. To compare the incidence of WSLs between conventional interdental cleaning tools with water floss among fixed appliance patients at T0, T1, T2, T3, and T4.
4. To see the correlation of oral plaque index (OPI) and WSLs between conventional interdental cleaning tools with water floss among fixed appliance patients at T0, T1, T2, T3, and T4.

Secondary Objectives

1. To see the effect of conventional interdental cleaning tools with water floss among fixed appliance patients on gingival health at T1, T2, T3 and T4.
2. To explore patients' perception of the usage of water flossers using self- administered questionnaires measured at T1 and T4.

Study design/Trial Design

The study will be designed based on the guidelines from the Consolidated Standards of Reporting Trials (CONSORT) statement and will be registered in Clinicaltrials.gov. All methods will be performed according to the relevant guidelines and regulations. The study was conducted according to the Declaration of Helsinki (as revised in 2013).

The study will be conducted in three phases:

i. Calibration of Orthodontic Plaque Index (OPI), Gingival Index (GI) and Enamel Decalcification Index (EDI) ii. Questionnaire translation and validation iii. Intervention: Baseline (T0, 0 months) and post-intervention (T1-T4, 3 to 12 months) The intervention study is a single-side blinded, two-arm parallel, prospective, single- centre randomised clinical trial. The study will be conducted from April 2024 to October 2025 in the Orthodontic Postgraduate Clinic, Universiti Malaya.

Participants

Participants will be recruited voluntarily based on inclusion and exclusion criteria; the centre would be located at the Orthodontic Postgraduate Clinic of Universiti Malaya. Informed and written consent will be obtained from the participants after the research procedure, and the research risks and benefits explained.

Inclusion and exclusion criteria:

Inclusion Criteria:

Mild to moderate crowding upper and lower arch 18 years old and above Patients with BPE score 0/1 Stay in areas with the same concentration of water fluoridation No history of orthodontic treatment before Able to read and understand in English or Bahasa Melayu Fit and healthy

Exclusion Criteria:

Severe crowding Less than 18 years old Patients with BPE score more than 2 Patients with systemic disease and syndromic Syndromic patients (eg; Cleft lip and palate) Unable to read and understand in English or Bahasa Melayu Clinically missing teeth (impacted/congenitally missing) Patients with upper and lower fixed appliance Patients with segmental fixed appliances in single or both arches.

Intervention In this research study, we would like to investigate incorporating water flossing into the oral hygiene routine, comparing it with oral hygiene practices with conventional interdental cleaning tools (Interdental brush and dental floss). The study design involves two groups: the intervention group, which will integrate water flossing into their daily oral care regimen, and the control group, which will adhere to their usual oral hygiene practices with conventional interdental cleaning tools.

Outcomes The study's outcomes will evaluate the presence and severity of white spot lesions through the Enamel Decalcification Index (EDI). Plaque accumulation will be assessed by employing the Orthodontic Plaque Index (OPI). Gingival health by using Gingival Index. A comprehensive questionnaire will be administered to determine the perceptions of interdental cleaning devices.

At Pre-Intervention (T0) : Full mouth scaling will be done and all study samples will be bonded with a straight-wire fixed appliance by the same bracket system McLaughlin, Bennett, and Trevisi (MBT) bracket system 022 x028 slot. Post-bond-up and diet instructions will be given to every participant.

Baseline data will be collected:

I.Orthodontic Plaque Index (OPI) Score 2.Gingival Index 3.Enamel decalcification index (EDI) score

Protocol for Orthodontic Plaque Index (OPI) data collection. The Orthodontic Plaque Index (OPI) will be conducted using a blunt probe with the scraping technique on the labial surfaces of teeth located mesial to the 6s. A disclosing tablet will not be utilised in this study due to its potential impact on the appearance of white spot lesions (WSLs).

Protocol for Gingival index A value is assigned to three tooth surfaces: vestibular, mesial, and distal. Lingual surfaces won't be included in our study. The periodontal probe is used with light pressure on the gingival sulcus to evaluate the bleeding. The assigned score to every surface is between 0 and 3 and it defines the level of gingival inflammation.

Protocol for Enamel Decalcification Index (EDI) data collection After the gingival assessment, the archwire and auxiliaries will be removed. Tooth surfaces will be cleaned using a slow-speed bristle brush without pumice, and the teeth will be dried before taking the intraoral images.

The primary investigator (ASAS) will take an intraoral clinical photo using a Canon EOS RP camera with an aperture of f/25, a shutter speed of 1/125, and an ISO of 500. A Godox ML-150 macro ring flash set at maximum intensity will be used for illumination. The images will be cropped and arranged using Canva.The Enamel Decalcification Index (EDI) representing the white spot lesions will be scored based on the Enamel Decalcification Index by (Banks & Richmond, 1994).

ELIGIBILITY:
Inclusion Criteria:

Mild to moderate crowding upper and lower arch 18 years old and above Patients with BPE score 0/1 Stay in areas with the same concentration of water fluoridation No history of orthodontic treatment before Able to read and understand in English or Bahasa Melayu Fit and healthy Patients with upper and lower fixed appliance

Exclusion Criteria:

Severe crowding Less than 18 years old Patients with BPE score more than 2 Patients with systemic disease and syndromic Syndromic patients (eg; Cleft lip and palate) Unable to read and understand in English or Bahasa Melayu Clinically missing teeth (impacted/congenitally missing) Patients with segmental fixed appliances in single or both arches.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
White spot lesion | From enrollment to the end of study at 8 months
  White spot lesion assessment using the Enamel Decalcification Index (EDI) by observing the clinical photos
Dental plaque | From enrollment to the end of study at 8 months
  Dental plaque using the Orthodontic Plaque Index (OPI)
Gingival health | From enrollment to the end of study at 8 months
  Gingival health assessment using the gingival index

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Universiti Malaya, Kuala Lumpur, Kuala Lumpur 50603, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patano A, Malcangi G, Sardano R, Mastrodonato A, Garofoli G, Mancini A, Inchingolo AD, Di Venere D, Inchingolo F, Dipalma G, Inchingolo AM. White Spots: Prevention in Orthodontics-Systematic Review of the Literature. Int J Environ Res Public Health. 2023 Apr 21;20(8):5608. doi: 10.3390/ijerph20085608. PMID 37107890
- [Background] Quaranta A, Marchisio O, D'isidoro O, Genovesi AM, Covani U. Single-blind randomized clinical trial on the efficacy of an interdental cleaning device in orthodontic patients. Minerva Stomatol. 2018 Aug;67(4):141-147. doi: 10.23736/S0026-4970.18.04104-3. Epub 2018 Feb 13. PMID 29495655
- [Background] Sarner B, Birkhed D, Andersson P, Lingstrom P. Recommendations by dental staff and use of toothpicks, dental floss and interdental brushes for approximal cleaning in an adult Swedish population. Oral Health Prev Dent. 2010;8(2):185-94. PMID 20589254
- [Background] Sawan N, Ben Gassem A, Alkhayyal F, Albakri A, Al-Muhareb N, Alsagob E. Effectiveness of Super Floss and Water Flosser in Plaque Removal for Patients Undergoing Orthodontic Treatment: A Randomized Controlled Trial. Int J Dent. 2022 Aug 31;2022:1344258. doi: 10.1155/2022/1344258. eCollection 2022. PMID 36090126
- [Background] Sharab L, Loss C, Jensen D, Kluemper GT, Alotaibi M, Nagaoka H. Prevalence of white spot lesions and gingival index during orthodontic treatment in an academic setting. Am J Orthod Dentofacial Orthop. 2023 Jun;163(6):835-842. doi: 10.1016/j.ajodo.2022.08.023. Epub 2023 Jan 29. PMID 36720655
- [Background] Smith AJ, Moretti AJ, Brame J, Wilder RS. Knowledge, attitudes and behaviours of patients regarding interdental deplaquing devices: A mixed-methods study. Int J Dent Hyg. 2019 Nov;17(4):369-380. doi: 10.1111/idh.12410. Epub 2019 Jun 27. PMID 31152632
- [Background] Sundararaj D, Venkatachalapathy S, Tandon A, Pereira A. Critical evaluation of incidence and prevalence of white spot lesions during fixed orthodontic appliance treatment: A meta-analysis. J Int Soc Prev Community Dent. 2015 Nov-Dec;5(6):433-9. doi: 10.4103/2231-0762.167719. PMID 26759794
- [Background] Vivaldi-Rodrigues G, Demito CF, Bowman SJ, Ramos AL. The effectiveness of a fluoride varnish in preventing the development of white spot lesions. World J Orthod. 2006 Summer;7(2):138-44. PMID 16779972
- [Background] Yazarloo S, Arab S, Mirhashemi AH, Gholamrezayi E. Systematic review of preventive and treatment measures regarding orthodontically induced white spot lesions. Dent Med Probl. 2023 Jul-Sep;60(3):527-535. doi: 10.17219/dmp/140964. PMID 37815515